CLINICAL TRIAL: NCT03665896
Title: A Comparison of Placement With the VivaSight Left-sided Double Lumen Tube With an Integrated Monitor/Camera Versus the Standard Left-sided Double Lumen Tube (DLT) With Fiberoptic Bronchoscopy in Patients Requiring One-lung Ventilation (OLV)
Brief Title: VivaSight Left-sided Double Lumen Tube Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Javier H Campos (Other)
Responsible Party: Sponsor-Investigator, Javier H Campos, Principle Investigator, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201302811
Record Dates: First submitted 2018-09-04; First posted 2018-09-11 (Actual); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Intubation, Intratracheal
Keywords: double-lumen endotracheal tube; VivaSight double-lumen tube
MeSH Terms: interventions — Intubation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VivaSight DLT group (Active Comparator): Thoracic surgery patient is intubated with VivaSight double-lumen tube (intubation with VivaSight double-lumen tube). The intubation time, duration between the passage of the tube through the vocal cords and the confirmation of proper tube positioning by the embedded camera, is recorded. The tube position is reconfirmed by fiberoptic bronchoscopy.
  Interventions: Device: intubation with VivaSight double-lumen tube; Procedure: fiberoptic bronchoscopy
- Standard DLT group (Placebo Comparator): Thoracic surgery patient is intubated with standard double-lumen tube (intubation with standard double-lumen tube). The intubation time, duration between the passage of the tube through the vocal cords and the confirmation of proper tube positioning by fiberoptic bronchoscopy, is recorded.
  Interventions: Device: intubation with standard double-lumen tube; Procedure: fiberoptic bronchoscopy

INTERVENTIONS:
Device: intubation with VivaSight double-lumen tube
  Arms: VivaSight DLT group
Device: intubation with standard double-lumen tube
  Arms: Standard DLT group
Procedure: fiberoptic bronchoscopy

SUMMARY:
The VivaSight™-DLT is a new OLV (one lung ventilation) device that contains an embedded camera. Therefore, a potential advantage is the continuous assessment of DLT position through continuous monitoring of the camera. The embedded camera of VivaSight™-DLT is positioned at the tracheal opening of the double lumen tube. It allows for continuous monitoring of the carina and bronchial tube placement.

The purpose of this study is to determine if a double lumen tube (DLT) with an embedded video camera, the VivaSight DLT, can be used in similar fashion to the standard double lumen tube with fiberoptic bronchoscopy. More specifically, the investigators would like to know the difference in time to optimal position in the left bronchus between the VivaSight DLT and the standard DLT with fiberoptic bronchoscopy. In addition, the investigators would like to know if the embedded camera on the VivaSight DLT provides a view that will allow for the optimum position of the DLT in the left bronchus.

DETAILED DESCRIPTION:
The investigators will perform a prospective, randomized study in thoracic surgical patients undergoing one-lung ventilation where the patient will receive either the VivaSight DLT or standard left-sided DLT. Subjects will be selected and evaluated who are at least 18 years old, but no older than 90 years old.

The investigators will compare the intubation time for the VivaSight™-DLT with the intubation time for standard DLT. The intubation time parameters for the VivaSight™-DLT are the passage of the tube through the vocal cords and the confirmation of proper tube positioning by the embedded camera. Fiberoptic bronchoscopy is performed to reassess the proper tube positioning, however, this will not be counted for the intubation time in this group. For the standard DLT, the intubation time parameter begins similarly, on the passage of the tube through the vocal cords, but ends with the confirmation of the proper placement by fiberoptic bronchoscopy. In both groups, C-MAC blade is used to visualize the passage of the tube through the vocal cords. These intubation times will be tracked real-time in the operating room and will be based upon both observation as well as the verbal confirmation of the attending anesthesiologist.

The intubation time must be within 5 minutes. The intubation time required more than 5 minutes is considered as unsuccessful intubation.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Adult patient undergoing scheduled thoracic surgery which requires double-lumen tube placement

Exclusion Criteria:

* More than 90 years of age
* Patients with emergency surgery
* Prisoners
* Patient who cannot provide their own consent
* Patient refusal
* Non-English speaking patients

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-07-10 (Actual); Primary Completion 2014-03-21 (Actual); Study Completion 2014-03-21 (Actual)

PRIMARY OUTCOMES:
Intubation time | Within 5 minutes
  We will compare the intubation time for the VivaSight double-lumen tube (DLT) with the intubation time for standard DLT.

SECONDARY OUTCOMES:
Picture reliability of the embedded camera of VivaSight double-lumen tube | Within 10 hours
  Picture reliability of the embedded camera will be assessed based upon the proper identification of the following structures; a) Carina, b) Left bronchial cuff , c) A radiopaque line of left bronchial tube, d) Right main bronchus.

CONTACTS AND LOCATIONS:
Overall Officials: Javier H Campos, MD, Principal Investigator — University of Iowa Hospitals & Clinics

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification will be shared with researchers who provide a methodologically sound proposal, to achieve aims in the approved proposal. IPD will be available for sharing immediately after publication and ending 5 years following article publication.
Supporting Information: Study Protocol
Time Frame: IPD will be available for sharing immediately after publication and ending 5 years following article publication.
Access Criteria: IPD will be accessible to researchers who provide a methodologically sound proposal, to achieve aims in the approved proposal.